CLINICAL TRIAL: NCT01344083
Title: Comparison of the Efficacy and Tolerability of T1210 and Olopatadine Hydrochloride 0.1% in the Treatment of Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LT1210-PII-04/10
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Seasonal Allergic Conjunctivitis
MeSH Terms: interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- T1210 (Experimental)
  Interventions: Drug: T1210
- Olopatadine hydrochloride (Active Comparator)
  Interventions: Drug: Olopatadine hydrochloride

INTERVENTIONS:
Drug: T1210 — 2 drops T1210 once a day
  Arms: T1210
Drug: Olopatadine hydrochloride — 2 drops once a day Olopatadine
  Arms: Olopatadine hydrochloride

SUMMARY:
The aim of this study is to compare the efficacy and the safety of T1210 versus Olopatadine eye drops in the topical treatment of seasonal allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Conjunctivitis allergic conjunctivitis

Exclusion Criteria:

* Severe ocular allergy
* Vernal keratoconjunctivitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the score of tearing | Day 28
Change from baseline of the score of itching | Day 28
Change from baseline of the score of conjunctival hyperaemia | Day 28

SECONDARY OUTCOMES:
Global local tolerance assessment by the Investigator and the patient | Day 7
Global local tolerance assessment by the Investigator and the patient | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Pierre Huguet, Clermont-Ferrand, France